CLINICAL TRIAL: NCT07322718
Title: A Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of the CD19-Targeting Circular RNA Product RXIM002 in Patients With Relapsed or Refractory B Cell-Mediated Autoimmune Diseases
Brief Title: Safety and Efficacy Study of RXIM002 in Severe, Relapsed or Refractory Autoimmune Diseases
Acronym: RXIM002
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: RiboX Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RX-AID-CS101
Record Dates: First submitted 2025-12-07; First posted 2026-01-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory B Cell-Mediated Autoimmune Diseases
Keywords: Autoimmune Disease
MeSH Terms: conditions — Recurrence; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RXIM002 (Experimental): Each study participant will be given 2 doses of RXIM002 at each dose level.
  Interventions: Biological: RXIM002 product

INTERVENTIONS:
Biological: RXIM002 product — Prior to infusion of the RXIM002 product, subjects will receive pre-medication if needed

SUMMARY:
This Phase 1, open-label study evaluates the safety, tolerability, and preliminary efficacy of RXIM002, a CD19-targeting circular RNA-mediated in-vivo CAR T-cell therapy, in adults with severe, relapsed, or refractory B cell-mediated autoimmune diseases.

DETAILED DESCRIPTION:
This Phase 1, open-label, single-arm, dose-escalation study is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary efficacy of RXIM002 in adults with severe, relapsed, or refractory B cell-mediated autoimmune diseases. Eligible participants will receive intravenous administration of RXIM002 and will be monitored for adverse events, laboratory parameters, and other safety outcomes. The study will also explore biological activity and potential clinical responses across the enrolled autoimmune conditions. Participants will be followed for a defined period after treatment to assess longer-term safety and durability of any observed effects. The study will include the following sequential phases: screening, treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntary agreement to provide written informed consent.
* Aged 18 to 65 years, either sex.
* Adequate organ function meeting screening criteria.
* Positive test for cluster of differentiation antigen 19 (CD19).

Systemic Lupus Erythematosus (SLE) and Lupus Nephritis (LN):

* Have been diagnosed with SLE or LN before screening.
* Presence of anti-dsDNA, anti-histone, anti-chromatin, anti-Ro (anti-SS-A), anti-La (anti-SS-B), antinuclear antibody (ANA), or anti-Sm antibodies at screening.
* Active disease at screening.
* Fulfill relapsed/refractory SLE or LN conditions

Lupus Nephritis (LN) :

* Kidney biopsy result indicating LN
* Evidence of LN disease activity

Systemic Sclerosis (SSc):

* Have been diagnosed with SSc before screening.
* Antinuclear Antibody (ANA) positive at screening or prior to screening. AND, evidence of SSc disease activity.
* Fulfill relapsed/refractory SSc conditions.

Immune Thrombocytopenia (ITP):

* Have been diagnosed with refractory ITP before screening.
* Platelet count <50×10⁹/L at screening.

Idiopathic Inflammatory Myopathy (IIM):

* Have been diagnosed with IIM before screening.
* Presence of at least 1 myositis specific (MSA), associated antibody (MAA), or ANA at screening or prior to screening.
* Evidence of IIM disease activity.
* Fulfill relapsed/refractory IIM conditions.

Membranous Nephropathy (MN):

* Have been diagnosed with MN before screening.
* Active MN patients meeting screening criteria.
* Fulfill relapsed/refractory MN conditions.

Autoimmune Hemolytic Anemia (AIHA):

* Have been diagnosed with AIHA before screening.
* Active AIHA patients meeting screening criteria.
* Fulfill relapsed/refractory AIHA conditions.

Exclusion Criteria:

* Active infections such as hepatitis and tuberculosis.
* Other autoimmune diseases.
* Serious underlying diseases such as active malignancies, uncontrolled diabetes.
* Female subjects who were pregnant, breastfeeding.
* Any uncontrolled psychiatric disorders (e.g., schizophrenia, bipolar disorder, eating disorders, major depression or anxiety disorder), as declared by the participant or reported in the medical records.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2027-12-19 (Estimated); Study Completion 2028-03-19 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Dose-Limiting Toxicities (DLTs) | 28 days after RXIM002 first infusion (Day 1)
Incidence and severity of treatment-emergent adverse events (TEAEs) | 52 weeks after RXIM002 first infusion (Day 1)
CAR positive cell Cmax | 24 weeks after RXIM002 first infusion (Day 1)
  CAR positive T cells in peripheral blood after RXIM002 infusion, maximum concentration (Cmax).
CAR positive cell Tmax | 24 weeks after RXIM002 first infusion (Day 1)
  CAR positive T cells levels in peripheral blood after RXIM002 infusion, time to Cmax (Tmax).
CAR positive cell AUC | 24 weeks after RXIM002 first infusion (Day 1)
  CAR positive T cells levels in peripheral blood after RXIM002 infusion, area under the concentration-time curve (AUC) .

SECONDARY OUTCOMES:
LNP (Lipid Nanoparticle) Cmax | 24 weeks after RXIM002 first infusion (Day 1)
  LNP in peripheral blood after RXIM002 infusion, maximum concentration (Cmax).
LNP (Lipid Nanoparticle) Tmax | 24 weeks after RXIM002 first infusion (Day 1)
  LNP levels in peripheral blood after RXIM002 infusion, time to Cmax (Tmax)
LNP (Lipid Nanoparticle) AUC | 24 weeks after RXIM002 first infusion (Day 1)
  LNP levels in peripheral blood after RXIM002 infusion, area under the concentration-time curve (AUC) .
CircleRNA Cmax | 24 weeks after RXIM002 first infusion (Day 1)
  CircleRNA in peripheral blood after RXIM002 infusion, maximum concentration (Cmax).
CircleRNA Tmax | 24 weeks after RXIM002 first infusion (Day 1)
  CircleRNA levels in peripheral blood after RXIM002 infusion, time to Cmax (Tmax).
CircleRNA AUC | 24 weeks after RXIM002 first infusion (Day 1)
  CircleRNA levels in peripheral blood after RXIM002 infusion, area under the concentration-time curve (AUC) .
Systemic Lupus Erythematosus (SLE) disease activity: Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | 52 weeks after RXIM002 first infusion (Day 1)
  Change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) scores from baseline up to 52 weeks, a total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
Systemic Sclerosis (SSc) disease activity :Modified rodnan skin score(mRSS) | 52 weeks after RXIM002 first infusion (Day 1)
  Change in modified Rodnan skin score (mRSS) from baseline up to 52 weeks in SSc patients. The mRSS is used to assess skin thickness and scope of SSc patients ,with a total score can fall between 0 and 51, with a higher score representing a more significant degree of skin involvement.
Idiopathic Inflammatory Myopathy (IIM) disease activity ：Manual muscle test-8 | 52 weeks after RXIM002 first infusion (Day 1)
  Change in manual muscle testing (MMT-8) score from baseline up to 52 weeks in IIM patients. This tool assesses muscle strength by testing 8 proximal, distal, and axial muscles ,assess unilateral(score range 0-80 points)handedness side, with a lower score representing a more significant degree of muscle involvement.
Autoimmune Hemolytic Anemia (AIHA) disease activity: Overall Hb therapeutic response | 8 weeks after RXIM002 first infusion (Day 1)
  At least one occurrence of Hb ≥ 100 g/L, concurrently with an increase of at least 20 g/L from baseline, and not attributable to red blood cell transfusion or other emergency therapeutic drugs
Immune Thrombocytopenia (ITP) disease activity: Overall response of platelet increment. | 8 weeks after RXIM002 first infusion (Day 1)
  The proportion of subjects whose platelet count recovered to ≥ 50 × 10^9/L and who did not require an increase in corticosteroid dose
Lupus Nephritis (LN) disease activity: Proportion of subjects achieving Primary Efficacy Renal Response(PERR) | 52 weeks after RXIM002 first infusion (Day 1)
  UPCR ≤ 0.7 g/g, with eGFR no more than 20% below the pre-lupus flare level or ≥ 60 mL/min/1.73 m², and no treatment failure event. Achieving Complete Renal Response (CRR)
Membranous Nephropathy (MN) disease activity: Clinical remission rate | 52 weeks after RXIM002 first infusion (Day 1)
  24-hour urinary protein quantification < 3.5 g/day with serum albumin > 30 g/L, and eGFR ≥ 85% of baseline value

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Huangpu District, China

IPD SHARING:
Plan to Share IPD: No